CLINICAL TRIAL: NCT04998786
Title: A Multi-center Open-label Phase 2 Study of Ixazomib, Iberdomide and Dexamethasone in Elderly Patients With Multiple Myeloma at First Relapse."
Acronym: I2D IFM2021_03
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC21_0169; 2021-001587-13 (EudraCT Number)
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma at First Relapse
Keywords: Multiple Myeloma, elderly patients, first relapse, previous exposed, High Risk, Ixazomib, Iberdomide, Dexametasone
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; iberdomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- assessment of treatment Ixazomib, dexamethasone, iberdomide (Experimental): Iberdomide, Ixazomib and Dexaméthasone during 6 cycles and Iberdomide and Ixazomib until progression
  Interventions: Drug: Ixazomib; Drug: Iberdomide; Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Ixazomib — Ixazomib 3 mg/day (days 1, 8, 15) cycle 1 to until progress
Drug: Iberdomide — Iberdomide 1.6 mg / day (day 1 to 21) cycle 1 to until progress
Drug: Dexamethasone Oral — Cycle 1 and 2 Dexaméthasone 20 mg/day on days 1, 8, 15, 22 Cycle 3 to 6 Dexamethasone 10 mg/day on days 1, 8, 15, 22

SUMMARY:
This is a phase II, multicenter, open-label study to evaluate the rate of patients achieving very good partial response (VGPR) or better to the oral combination Iberdomide Ixazomib Dexamethasone in elderly patients with multiple myeloma at first relapse .

The patient population will consist of adult men and women more than 70 years, who meet eligibility criteria.

Following the screening period, patients will be enrolled and treated then, they will receive therapy with Iberdomide, Ixazomib and Dexaméthasone during 6 cycles and Iberdomide and Ixazomib until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 70 years
2. Eastern Collaborative Oncology Group (ECOG) performance score of ≤2
3. Life expectancy > 6 months
4. Voluntary written informed consent must be given before performance of any study-related procedure not part of normal medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
5. Symptomatic multiple myeloma (MM) at first relapse, as defined below:

   * Symptomatic multiple myeloma according to international criteria.(Rajkumar et al, 2014)
   * Relapsed MM is defined as previously treated MM that progresses and requires initiation of salvage therapy.
6. Subject must have received one prior line of therapy for at least 3 cycles.
7. Subject has measurable disease at Screening, defined at least one of the following:

   * Serum M-protein ≥ 0.5 gram (g)/deciliter (dL), OR
   * Urine M-protein ≥ 200 mg in 24 hours, OR
   * Serum immunoglobulin free light chain (FLC) ≥ 10 mg/dL provided serum FLC ratio is abnormal.
8. Subjects must meet the following laboratory parameters, per laboratory reference range (performed at most 15 days before cycle 1 day 1):

   * Absolute neutrophil count (ANC) ≥ 1000/microliter (μL). Subjects may use growth factor support to achieve ANC eligibility criteria.
   * Platelet count ≥ 75,000 /mm3 for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count ≥ 50,000/mm3 for subjects in whom > 50% of bone marrow nucleated cells are plasma cells. It is not permissible to transfuse subjects to achieve minimum platelet counts within 3 days before study.

     --AST and ALT ≤ 3 × upper limit of normal (ULN).
   * Total bilirubin ≤ 1.5 × ULN. Subjects with documented Gilbert's syndrome may have bilirubin > 1.5 × ULN with the approval of the Primary Therapeutic Area Medical Director
   * Creatinine clearance (CrCl) ≥ 30 milliliter (mL)/minute (min) (using Cockroft and Gault Formula)
9. Patient should comply with Celgene's pregnancy prevention plan for Iberdomide (please see appendix 8 Iberdomide Pregnancy Prevention Plan for subjects in clinical trials)
10. Female patients who:

    * are postmenopausal for at least 24 months before the screnning visit, OR
    * are surgically sterile (have undergone a hysterectomy or bilateral oophorectomy)
11. Men even if surgically sterilized must agree to not father a child and agree to practice complete abstinence or to use a condom during therapy and dose interruptions and for 90 days after the last dose of study drug, even if they have had a successful vasectomy, if their partner is of childbearing potential or pregnant.

Non-inclusion Criteria:

1. Subject is refractory to bortezomib, defined as progression on or within 60 days of the last dose of bortezomib.
2. Subject has had prior treatment with ixazomib, carfilzomib, pomalidomide or iberdomide
3. Subject has any of the following conditions:

   * Non-secretory or oligo-secretory MM
   * Light chain Amyloidosis (AL Amyloidosis)
   * POEMS syndrome Waldenström macroglobulinemia
4. Known Human Immunodeficiency Viral (HIV) infection
5. Active hepatitis B or C infection based on blood screen tests
6. Significant cardiovascular or pericardial disease, including uncontrolled angina, hypertension, arrhythmia, recent myocardial infarction within 6 months, congestive, heart failure New York Heart Association (NYHA) Class ≥ 3
7. Major surgery within 4 weeks prior screening
8. Acute infections requiring parenteral therapy (antibiotic, antifungal or antiviral) within 14 days
9. ≥ Grade 3 Peripheral neuropathy or grade 2 with pain
10. Uncontrolled diabetes or uncontrolled hypertension within 14 days
11. Any other medical condition that, in the opinion of the Investigator, would adversely affect the subject's participation in the study
12. Subject has a history of other active malignancies, including myelodysplastic syndrome (MDS), within the past 3 years prior to study entry, with the following exceptions:

    * Adequately treated in situ carcinoma of the cervix uteri or the breast,
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin,
    * Prostate cancer Gleason grade 6 or lower AND with stable Prostate Specific Antigen (PSA) levels off treatment,
    * Previous malignancy with no evidence of disease confined and surgically resected (or treated with other modalities) with curative intent and unlikely to impact survival during the duration of the study.
13. Known intolerance to steroid therapy
14. Serious medical or psychiatric illness likely to interfere with participation in study
15. Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs
16. Subjects unable or unwilling to undergo antithrombotic prophylactic treatment
17. Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients have very good partial response (VGPR) or better | approximate 18 months
  Using IMWG criteria

SECONDARY OUTCOMES:
Number of adverse events | approximate 18 months
  Number of adverse events defined by Common Terminology Criteria for Adverse Events (v5)
Number of responses | 3 months
  Partial Response (PR), Very Good Partial Response (VGPR), Complete Response (CR) and minor response (MR) will be evaluated according to IMWG
Number of responses | 6 months
  Partial Response (PR), Very Good Partial Response (VGPR), Complete Response (CR) and minor response (MR) will be evaluated according to IMWG
Number of the death | approximate 18 months
  is defined as the time in months from inclusion to the date of death due to any cause. Subject alive will be censored at the last known alive date.
Number of progression | approximate 18 months
  is defined as the time in months from inclusion to the date of disease progression or death due to any cause, using IMWG criteria
Percentage of time to progression | approximative 18 months
  is defined as the time in months from inclusion to the date of disease progression or death due to any cause, using IMWG criteria
Percentage of duration of response | approximative 18 months
  is defined as the time from the first response (PR or better) to the date of disease progression or death due to any cause
Percentage of duration of therapy | approximative 18 months
  is defined as the time from treatment initiation to the last dose of therapy
Percentage of time to response | approximative 18 months
  according IMWG
Percentage of Overall Response Rate | approximative 18 months
  according IMWG
Percentage of value of biological prognostic factors | day 1
  prognostic factors as ISS stage, cytogenetic as del(17p), t(4;14),
Percentage of frailty scores | day 1
  age, ECOG, comorbidity index
Percentage of score of quality of life | approximative 18 months
  To assess Quality of Life EQ5D and SF36

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Touzeau, Principal Investigator — Nantes University Hospital
Locations (21):
- France (21):
  - CHR, Annecy
  - CH de la cote basque, Bayonne
  - CHRU Hopital Haut Lévêque, Bordeaux
  - CHU, Caen
  - CHU, Clermont-Ferrand
  - CHRU, Dijon
  - CHD les Oudairies, La Roche-sur-Yon
  - CHRU Lille, Lille
  - CHU, Limoges
  - CH Lyon Sud, Lyon
  - CHRU, Nancy
  - CHU, Nantes
  - Hopital de l'archet, Nice
  - CHU Henri Mondor, Paris
  - Hopital St Antoine, Paris
  - Hôpital Cochin, Paris
  - University Hospital, Poitiers
  - CHRU, Rennes
  - ICANS, Strasbourg
  - CHU, Toulouse
  - CHRU Bretonneau, Tours